CLINICAL TRIAL: NCT05228041
Title: Real Life Assessment of Biologics Efficacy in Severe Chronic Rhinosinusitis With Nasal Polyps
Brief Title: BIOlogics in Severe Nasal POlyposis SurvEy
Acronym: BIOPOSE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: DRI_2021/0030
Record Dates: First submitted 2021-12-17; First posted 2022-02-08 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Biologic; nasal polyp; chronic rhinosinusitis; eosinophil; endotype
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab; mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Biologic treatments available in CRSwNP (dupilumab, mepolizumab and benralizumab according to their marketing approval) — Drug prescription according to their marketing approval (subcutaneously, every month or every two weeks)

SUMMARY:
With a prevalence of 2-4% in western countries, Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) is of major concern regarding its substantial impact on the social and physical quality of life. So far, endoscopic sinus surgery remains the treatment of choice when the first line of medical treatment with corticosteroid has failed.

During the last 15 years, several studies have shown that CRSwNP is associated with a T helper 2 (T2) immune response leading to B cell release of IgE, mucosal recruitment of eosinophils from bone marrow via Interleukin (IL)-5, IL-4 and IL-13 mediated chemoattractant production.

New biologic agents capable of blocking T2 cytokines have been developed in the field of eosinophil-associated diseases, shifting the paradigm of treatment for patients with CRSwNP. In the near future, endotype profiling with accurate biomarkers will be mandatory to tailor the treatment of nasal polyposis with specific biologic therapies.

Herein we propose a prospective study monitoring medical records of CRSwNP patients who undergo biologic treatments. The objectives are to assess treatment efficacy on quality of life, to report clinical and biological criteria for prescription and to measure tolerance and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients of over 18-year old requiring a biologic treatment for CRswNP in accordance with its marketing approval

Exclusion Criteria:

* Oral corticotherapy in the previous month;
* Biologic treatment with anti-IgE (omalizumab), anti-IL-5/IL-5R (mepolizumab, benralizumab) or anti-IL-4/IL-13R (dupilumab) or any other biotherapy for inflammatory diseases in the previous 6 months apart from ongoing biotherapies for severe asthma;
* Hypersensitivity to humanized antibodies ;
* Documented SARS-Cov2 infection in the last 3 months with persistent olfactory disorders related to COVID;
* Pregnant or breast-feeding women;
* Patient without social coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of over 18-year old requiring a biologic treatment for CRswNP in accordance with its marketing approval
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
6-month rate of patients with a SNOT-22 (Sinonasal Outcome test -22) score change over the minimal clinically important difference of 8.9 by comparison of SNOT-22 scores measured at Month 0 and Month 6 | Day0, Month 6
  from 0 to 110 , 110 = worst outcome

SECONDARY OUTCOMES:
SNOT 22 (Sinonasal Outcome Test-22) scores | Day 0, Month 3, Month 6, Month 12 and Month 18
  from 0 to 110 , 110 = worst outcome
Visual analogical scale (VAS) for nasal obstruction | Day 0, Month 3, Month 6, Month 12 and Month 18
  from 0 to 10, 10 = worst outcome
Visual analogical scale (VAS) for smell lost | Day 0, Month 3, Month 6, Month 12 and Month 18
  from 0 to 10, 10 = worst outcome
Visual analogical scale (VAS) for rhinorrhea | Day 0, Month 3, Month 6, Month 12 and Month 18
  from 0 to 10, 10 = worst outcome
Visual analogical scale (VAS) for craniofacial pain | Day 0, Month 3, Month 6, Month 12 and Month 18
  from 0 to 10, 10 = worst outcome
Number of systemic corticosteroid treatment courses between each visit | Day 0, Month 3, Month 6, Month 12 and Month 18
Delay to first surgical procedure | Day 0, Month 3, Month 6, Month 12 and Month 18
Blood eosinophil count | Day 0, Month 3, Month 6, Month 12 and Month 18
  number of cells per mm3
Blood total IgE concentrations | Day 0, Month 3, Month 6, Month 12 and Month 18
  concentration expressed by KUI/L

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Mortuaire, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France

REFERENCES:
- [Derived] Favier V, Daveau C, Carsuzaa F, Fieux M, Vandersteen C, Castillo L, Papon JF, de Gabory L, Saroul N, Verillaud B, Rumeau C, Jankowski R, Michel J, de Bonnecaze G, Lecanu JB, Coste A, Bequignon E, Malard O, Mortuaire G. Study protocol: the biologics in severe chronic rhinosinusitis with nasal polyps survey. BMJ Open. 2024 May 15;14(5):e083112. doi: 10.1136/bmjopen-2023-083112. PMID 38749694